CLINICAL TRIAL: NCT05948228
Title: Principal Investigator,Resident at Cairo University
Brief Title: Prevention of White Spot Lesions Using Bioactive Gel
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farah Khaled El Hindawy, Prevention of white spot lesions in patients undergoing orthodontic treatment using bioactive gel versus fluoride gel, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Giomer based bioactive gel
Record Dates: First submitted 2023-06-24; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: White Spot Lesions
Keywords: white spot lesions; orthodontic treatment; Prevention; bioactive gel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of bioactive gel on teeth in patients assigned for orthodontic treatment (Experimental): Application of bioactive gel on labial/buccal surfaces of teeth is done according to manufacturer instructions using microbrush followed by light curing
  Interventions: Drug: giomer based bioactive gel
- Application of Fluoride on teeth in patients assigned for orthodontic treatment (Active Comparator): Application of fluoride gel will be done using a gel loaded tray held in the mouth for 4 minutes .After removal of tray ,patients must spit out the residual gel. The use of suction is a must to avoid the problem of over ingestion
  Interventions: Drug: Fluoride gel

INTERVENTIONS:
Drug: giomer based bioactive gel — Application of bioactive gel to prevent white spot lesions in orthodontic patients
  Arms: Application of bioactive gel on teeth in patients assigned for orthodontic treatment
Drug: Fluoride gel — Application of fluoride gel to prevent white spot lesions in orthodontic patients
  Arms: Application of Fluoride on teeth in patients assigned for orthodontic treatment

SUMMARY:
white spot lesions are a common problem and are reported in up to 96% of orthodontic patients. In this study, the preventive effect of bioactive gel is evaluated in comparison to fluoride.

DETAILED DESCRIPTION:
Dental caries is a chronic infectious disease present worldwide and is among one of the most common oral diseases. It is a multifactorial disease resulting from imbalance between demineralization and remineralization initiated by acid producing bacteria in the microenvironment.

The incipient form of caries, white spot lesions (WSL), is characterized by primitive enamel surface and subsurface demineralization and could be identified clinically by their chalky white appearance . Orthodontic treatment is a major risk factor for the development of WSL. They are reported in up to 96% of orthodontic patients.

Many materials are being used to prevent white spot lesions with fluoride being the most commonly used . New materials have been emerged such as giomer based bioactive gel with the ability to release six ions Fluoride inhibits demineralization and promotes deposition of fluoroapatite. Aluminum helps to decrease demineralization as well by forming Alumino fluoro complexes. Borate reduces biofilm formation beside its antibacterial effect.

Silica promotes remineralization by inducing apatite nucleation on the tooth surface. Strontium converts hydroxyapatite into strontium apatite thus increasing acid resistance and has an inhibitory effect on bacterial growth. Other ions such as Na act as strong base and have acid buffer capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned for orthodontic treatment with fixed appliances
* Sound teeth with fixed orthodontic appliances
* Either maxillary or mandibular teeth or both

Exclusion Criteria:

* Patients with poor oral hygiene
* Allergic reaction to the materials used.
* Lack of compliance.
* xerostomia
* Evidence of parafunctional habits.
* Active carious lesions
* Dental fluorosis
* Hypocalcified teeth
* Systemic diseases affecting teeth such as Amelogenesis imperfecta
* Severe periodontal affection

Ages: 15 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
incidence of white spot lesions using DIAGNOdent | Baseline,change from baseline at 3 months,6 months,9 months and 12 months
  the ability of the gels to prevent white spot lesions will be assessed using DIAGNOdent

SECONDARY OUTCOMES:
incidence of white spot lesions using ICDAS (international caries detection and assessment system) | Baseline,change from baseline at 3 months,6 months,9 months and 12 months
  the ability of the gels to prevent white spot lesions will be assessed using ICDAS